CLINICAL TRIAL: NCT01741025
Title: A Multicenter Randomized Controlled Post-market Clinical Follow-up Trial Comparing the Effectiveness and Safety of the iFuse Implant System® Versus Conservative Management for Patients With Chronic, Disabling SI Joint Pain.
Brief Title: iFuse Implant System® Minimally Invasive Arthrodesis
Acronym: iMIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 300134
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Sacroiliac Joint Pain
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iFuse Implant System (Experimental): Surgical placement of iFuse implants in the affected SI joint
  Interventions: Device: iFuse Implant System
- conservative management (Active Comparator): Medications, physical therapy, information
  Interventions: Other: Conservative Management

INTERVENTIONS:
Device: iFuse Implant System — Placement of iFuse implant system via surgery
  Arms: iFuse Implant System
Other: Conservative Management — Medications for pain, physical therapy, cognitive behavour therapy
  Arms: conservative management

SUMMARY:
The purpose of this study is to compare outcomes when patients with chronic sacroiliac joint pain undergo either SI joint fusion with the iFuse Implant System or undergo conservative management of the SI joint

DETAILED DESCRIPTION:
This study is a multicenter randomized controlled, post-market clinical follow-up clinical trial of the iFuse Implant System for SI joint fusion vs. conservative management. Subjects assigned to conservative management may cross over to iFuse after a minimum of 6 months of conservative treatment. Conservative management does not include interventional procedures such as prolotherapy, steroid injections and/or RF ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-70 at time of screening
2. Patient has lower back pain for >6 months or >18 months for pregnancy induced lower back pain
3. Diagnosis of the SI joint as the primary lower back pain generator based on ALL of the following: a. Patient has pain at or close to the posterior superior iliac spine (PSIS) with possible radiation into buttocks, posterior thigh or groin and can point with a single finger to the location of pain (Fortin Finger Test), and b. Patient has at least 3 of 5 physical examination maneuvers specific for SI joint pain, and c. Patient has improvement in lower back pain NRS of at least 50% of the pre injection NRS score after fluoroscopic controlled injection of local anesthetic into affected SI joint(s) (including previous documented test <6 months ago)
4. Baseline Oswestry Disability Index (ODI) score of at least 30%
5. Baseline lower back pain score of at least 50 on 0-100 point VAS
6. Patient has signed study-specific informed consent form
7. Patient has the necessary mental capacity to participate and is physically able to comply with study protocol requirements

Exclusion Criteria:

1. Severe lower back pain due to other causes, such as lumbar disc degeneration, lumbar disc herniation, lumbar spondylolisthesis, lumbar spinal stenosis, lumbar facet degeneration, and lumbar vertebral body fracture
2. Sacroiliac pathology caused by auto-immune disease (e.g. ankylosing spondylitis) and/or neoplasia (e.g. benign or malignant tumor) and/or crystal arthropathy
3. History of recent (<1 year) fracture of the pelvis with documented malunion, non-union of sacrum or ilium or any type of internal fixation of the pelvic ring.
4. Spine surgery during the past 12 months.
5. Previously diagnosed or suspected osteoporosis (defined as prior T-score <-2.5 or history of osteoporotic fracture)
6. Documented osteomalacia or other metabolic bone disease
7. Any condition or anatomy that makes treatment with the iFuse Implant System infeasible
8. Known allergy to titanium or titanium alloys
9. Use of medications known to have detrimental effects on bone quality and soft-tissue healing
10. Prominent neurologic condition that would interfere with physical therapy
11. Current systemic infection or local infection at the SI joint
12. Currently pregnant or planning pregnancy in the next year
13. Known or suspected drug or alcohol abuse
14. Diagnosed psychiatric disease (e.g., schizophrenia, major depression, personality disorders) that could interfere with study participation
15. Patient is participating in an investigational study or has been involved in an investigational study within 3 months of surgery

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12-15 (Actual); Study Completion 2017-09-24 (Actual)

PRIMARY OUTCOMES:
The change in lower back pain as rated by the study subject using a 0-100 visual analog scale (VAS) at 6 months after initiation of treatment | 6 months

SECONDARY OUTCOMES:
Change from baseline in lower back pain (VAS) | 1, 3, 12 and 24 months
Change from baseline in leg pain (VAS | 1, 3, 6, 12 and 24 months
Change in disability due to back pain (ODI | 3, 6, 12 and 24 months
Change in quality of life (EQ-5D | 3, 6, 12 and 24 months
Change in ambulatory and work status | 1, 3, 6, 12 and 24 months
Change in depression score (Zung Depression Scale | 3, 6, 12 and 24 months
Change in objective functional test (ASLR | 3, 6, 12 and 24 months
Change in walking distance | 3, 6, 12 and 24 months
Patient satisfaction and self-rating of disease state | 3, 6, 12 and 24 months
Serious adverse events | during 24 months
Device breakage, loosening and migration | 12 months

OTHER OUTCOMES:
Surgical re-interventions of target SI joint(s) | over 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cher, Study Director — SI-BONE, Inc.
Locations (9):
- Belgium (2):
  - OLV Ziekenhuis Aalst, Aalst
  - La Clinique de l'Espérance, Montegnée
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Praxisgemeinschaft "Leben in Bewegung", Hilden
- Italy (3):
  - Istituto Ortopedico Rizzoli, Bologna
  - Ospedale Civile Di Legnano, Legnano
  - IRCCS Policlinico San Matteo, Pavia
- Aleris Specialistvård Ängelholm, Ortopedkliniken, Ängelholm, Sweden

REFERENCES:
- [Derived] Dat KO, Cher D, Polly DW. Effects of BMI on SI joint fusion outcomes: examining the evidence to improve insurance guidelines. Spine J. 2024 May;24(5):783-790. doi: 10.1016/j.spinee.2023.11.015. Epub 2023 Dec 9. PMID 38081463
- [Derived] Dengler JD, Kools D, Pflugmacher R, Gasbarrini A, Prestamburgo D, Gaetani P, van Eeckhoven E, Cher D, Sturesson B. 1-Year Results of a Randomized Controlled Trial of Conservative Management vs. Minimally Invasive Surgical Treatment for Sacroiliac Joint Pain. Pain Physician. 2017 Sep;20(6):537-550. PMID 28934785
- [Derived] Dengler J, Sturesson B, Kools D, Prestamburgo D, Cher D, van Eeckhoven E, Erk E, Pflugmacher R, Vajkoczy P; the iMIA study group. Referred leg pain originating from the sacroiliac joint: 6-month outcomes from the prospective randomized controlled iMIA trial. Acta Neurochir (Wien). 2016 Nov;158(11):2219-2224. doi: 10.1007/s00701-016-2953-7. Epub 2016 Sep 15. PMID 27629371
- [Derived] Sturesson B, Kools D, Pflugmacher R, Gasbarrini A, Prestamburgo D, Dengler J. Six-month outcomes from a randomized controlled trial of minimally invasive SI joint fusion with triangular titanium implants vs conservative management. Eur Spine J. 2017 Mar;26(3):708-719. doi: 10.1007/s00586-016-4599-9. Epub 2016 May 14. PMID 27179664
- Available data/document: publication 6 month results — https://www.ncbi.nlm.nih.gov/pubmed/27179664
- Available data/document: publication 6 month results — https://www.ncbi.nlm.nih.gov/pubmed/27629371